CLINICAL TRIAL: NCT01513668
Title: An Open Label, Balanced, Randomised, Two-treatment, Two-period, Two-sequence, Single Dose, Crossover Bioavailability Study Comparing Acetaminophen 650 mg Extended Release Gel Tabs (Containing Acetaminophen 650 mg) of OHM Laboratories (Subsidiary of Ranbaxy) With Tylenol 8 Hour 650 mg Gel Tabs (Containing Acetaminophen 650 mg) of Mc Neil, Consumer & Speciality Pharmaceuticals in Healthy, Adult, Human, Male Subjects Under Fed Condition
Brief Title: A Relative Bioavailability Study of Acetaminophen Extended Release Gel Tabs 650 mg Under Fed Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Sponsor
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 202_ACETA_06
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetaminophen extended release Gel tabs (Experimental): Acetaminophen extended release Gel tabs 650 mg of OHM Laboratories Inc. (A subsidiary of Ranbaxy Pharmaceuticals Inc., USA)
  Interventions: Drug: Acetaminophen
- Tylenol® 650 mg (Active Comparator): Tylenol® 650 mg of McNeil Consumer and Specialty Pharmaceuticals, Division of McNeil PPC, INC. Fort Washington, PA 19034 USA
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — Extended release Gel tabs 650 mg

SUMMARY:
The purpose of this study is to compare single-dose oral bioavailability of acetaminophen 650 mg extended release geltabs (containing acetaminophen 650 mg) of OHM Laboratories, USA (subsidiary of Ranbaxy) with Tylenol extended release geltabs (containing acetaminophen 650 mg) of Mc Neil, Consumer & Specialty Pharmaceuticals, U.S.A in healthy, adult, male human subjects under fed condition.

DETAILED DESCRIPTION:
The study was conducted as open label, balanced, randomised, two-treatment, two-period, two-sequence, single dose, crossover bioavailability study comparing acetaminophen 650 mg extended release gel tabs (containing acetaminophen 650 mg) of OHM Laboratories (subsidiary of Ranbaxy) with Tylenol 8 Hour 650 mg extended release gel tabs (containing acetaminophen 650 mg) of Mc Neil, Consumer & Specialty Pharmaceuticals in healthy, adult, human, male subjects under fed condition.

The treatments were assigned to the study subjects according to SAS generated randomization schedule. Each subject received a single oral dose either Test or Reference product in each period with 240ml of water at ambient temperature, 30 minutes after start of a high-fat high calorie breakfast during each period of the study under supervision of a trained medical officer.

During the course of study, the safety parameters including vital signs, physical examination, medical history, clinical laboratory and safety tests (haematology, biochemical parameters) were assessed and clinical laboratory safety tests (hematology & biochemical parameters) were performed again at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

Aged 18-45 years.

* Had a non-vegetarian diet.
* Were neither overweight nor underweight for their height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
* Had voluntarily given written informed consent to participate in this study.
* Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.

Exclusion Criteria:

* Had history of hypersensitivity to acetaminophen or to any of the components of the formulation.
* Had any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
* Had presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
* Had presence of values that were significantly different from normal reference ranges and/or judged clinically significant for haemoglobin, total white blood cells count, differential WBC count or platelet count.
* Were positive for urinary screen testing of drugs of abuse (opiates or cannabinoids).
* Had presence of values, which were significantly different from normal reference ranges and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
* Had clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), glucose (positive) or protein (positive).
* Had clinically abnormal ECG or Chest X-ray.
* Had history of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or hematological disease, diabetes or glaucoma (rise of pressure inside the eye leading to blurring or loss of vision).
* Had history of any psychiatric illness, which may impair the ability to provide written informed consent.
* Were regular smokers who smoked more than 10 cigarettes daily or had difficulty abstaining from smoking for the duration of each study period.
* Had history of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or had difficulty in abstaining for the duration of each study period.
* Had used any enzyme modifying drugs within 30 days prior to Day 1 of this study.
* Had participated in any clinical trial within 12 weeks preceding Day 1 of this study.
* Subjects who, through completion of this study, had donated and/or lost more than 350 mL of blood in the past 3 months.

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-05; Primary Completion 2006-05 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) and Peak Plasma Concentration (Cmax) of Acetaminophen | 0 to 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology Unit, B-22, Sector 62, Noida, Uttar Pradesh, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html